CLINICAL TRIAL: NCT06536686
Title: Silent Myocardial Ischemia in Patients Undergoing Non-oncological Abdominal Surgeries
Status: Recruiting | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: 7/2024
Record Dates: First submitted 2024-07-24; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Silent Myocardial Ischemia; Acute Myocardial Infarction
Keywords: acute coronary syndrome; silent myocardial ischemia; troponin T; NT-pro BNP; genetic polymorphisms; miRNA; extracellular vesicles
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The first group- silent myocardial ischemia
  Interventions: Genetic: Silent myocardial ischemia, STEMI
- The second group -STEMI undergoing primary coronary angiography.
  Interventions: Genetic: Silent myocardial ischemia, STEMI

INTERVENTIONS:
Genetic: Silent myocardial ischemia, STEMI — Silent myocardial ischemia association with genetic polymorphisms, miRNA and EVs

SUMMARY:
Perioperative mortality in non-cardiac surgical procedures is 1-2 % with half of these cases attributed to cardiovascular events. Silent myocardial ischemia, which typically occurs within 72 hours to 30 days after surgery is the most common. The only diagnostic criterion is troponin T, which should ideally be measured before the operation. In addition to troponin, blood samples can be taken for N terminal-pro BNP. Genetic factors can also contribute to the development of myocardial infarction. Methylenetetrahydrofolate reductase (MTHFR) is an important enzyme in homocysteine metabolism. The two most investigated variants of the MTHFR gene are C677T and A1298C single nucleotide polymorphisms (SNPs). As new biomarkers of cardiovascular diseases, non-coding RNAs, especially microRNAs (miRNAs) and circulating extracellular vesicles (EVs) are of interest. On the other hand, EVs were shown to reduce myocardial autophagy, leading to death during MI or ischemic-reperfusion injury. Methods: The investigators will enroll approximately 200 patients aged 18 and older. The first study of silent myocardial ischemia, will include patients without cardiovascular disease undergoing urgent or elective surgery for benign abdominal diseases. The second group will include patients with STEMI undergoing primary coronary angiography. Patients will also complete a questionnaire on folate intake. Subsequently, the investigators will collect blood for standard laboratory tests as well as troponin T, N terminal-pro BNP, homocysteine, and folic acid. Blood will be also collected for biomarker analysis. On the third day of hospitalization, blood will be collected again for troponin T, NT-proBNP and biomarkers. After that, the investigators will follow up the patients for another year every three months for the possible occurrence of major adverse cardiovascular events (MACE). Peripheral blood and blood from the coronary sinus will be collected in patients from the second study group for biomarker research. Expected results and significance for science and medicine: the investigators anticipate that the study will improve the understanding of clinical, biochemical, and biological markers of silent ischemia and cardiovascular complications following non-oncological abdominal surgeries. Knowledge of these factors would enable early identification of patients at higher risk of such complications, leading to more targeted preoperative preparation for non-oncological abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-oncological abdominal disease and without cardiovascular disease
* Patients with STEMI

Exclusion Criteria:

* Patients with active cancer
* Pregnant women
* Psychiatric patients
* Patient with dementia
* Patients who do not understand basic instructions
* Alcohol and illegal drug addicts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the first group we will enroll 100 patients aged 18 and older without cardiovascular disease, which will undergo treatment for non-oncological abdominal procedures. Upon admission, they will complete a questionnaire regarding folate intake from food. We will follow all patients for 72 hours post-surgery and then for an additional 12 months , with telephone follow-ups every 3 months. We will record data on whether they experienced MACE during this period. Blood samples, such as troponin T and NT-proBNP, hsCRP, lipid profile, homocysteine, folic acid, and samples for biological markers, will be collected immediately upon admission. On the third day, blood will be collected for troponin T and NT-proBNP and biomarkers. In second group, we will recruit 100 patients with STEMI for PCI.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of silent ischemia | 12 months
  To investigate the incidence of silent ischemia in a group of patients hospitalized because of acute and chronic non-oncological abdominal surgery.
Incidence of MACE | 12 months
  To investigate the incidence of major adverse cardiovascular events (MACE) within a one year from the discharge from the hospital
Association with genetic polymorphisms | 1 month
  To investigate the association of folate pathway genetic polymorphisms with silent ischemia
Association with miRNA | 1 month
  To investigate the role of miRNAs as biomarkers in silent ischemia
Association with EVs | 1 month
  To investigate the role of EVs as biological markers in silent ischemia
STEMI and biomarkers | 1 month
  To validate the presence of the candidate biomarkers in STEMI

CONTACTS AND LOCATIONS:
Overall Officials: Jasna Klen, MD, PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No